CLINICAL TRIAL: NCT05883488
Title: Effectiveness of Robot-Assisted Upper Extremity Rehabilitation in Children With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AnkaraCHBilkent-BT
Record Dates: First submitted 2023-03-13; First posted 2023-06-01 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-05

CONDITIONS: Cerebral Palsy; Upper Extremity Problem
Keywords: Cerebral Palsy; Robotic rehabilitation; Upper extremity
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic rehabilitation group (Experimental): The robotic rehabilitation group will receive a robot-assisted upper extremity rehabilitation program in addition to the conventional rehabilitation program.The robotic rehabilitation program (with the Armeo Spring Pediatric Robotic Rehabilitation system) will be implemented 3 days a week for 30 minutes.
  Interventions: Other: Robot-assisted upper extremity rehabilitation; Other: Conventional rehabilitation
- Conventional rehabilitation group (Active Comparator): Conventional rehabilitation program will be applied 5 days a week, lasting 60 minutes.
  Interventions: Other: Conventional rehabilitation

INTERVENTIONS:
Other: Robot-assisted upper extremity rehabilitation — The robotic rehabilitation program (with the Armeo Spring Pediatric Robotic Rehabilitation system) will be implemented 3 days a week for 30 minutes in addition to the conventional rehabilitation program. Participants will receive a total of 4 weeks of treatment.
  Arms: Robotic rehabilitation group
Other: Conventional rehabilitation — Conventional rehabilitation program will be applied 5 days a week, lasting 60 minutes.

SUMMARY:
The use of robotic rehabilitation, a treatment method for improving the motor functions of the upper extremities, is gradually increasing in children with cerebral palsy.

The aim of this study is to investigate the effect of robot-assisted rehabilitation for the upper extremity on upper extremity functions, manual skills and quality of life in patients with unilateral or bilateral/triplegic spastic cerebral palsy and also to compare the effect of robot-assisted upper extremity rehabilitation compared to traditional rehabilitation methods.

DETAILED DESCRIPTION:
In this study, it was planned to include 42 patients diagnosed with unilateral or bilateral/triplegic spastic cerebral palsy, aged 5-15 years, who were treated in the Pediatric Rehabilitation Service of Ankara City Hospital Physical Therapy and Rehabilitation Hospital, and met the inclusion criteria.

Participants will be divided into two groups as study and control groups. In addition to the conventional rehabilitation program, the study group will be included in the robot-assisted upper extremity rehabilitation program, while the control group will be included in the conventional rehabilitation program only.

Conventional rehabilitation program will be applied 5 days a week, lasting 60 minutes. The robotic rehabilitation program (with the Armeo Spring Pediatric Robotic Rehabilitation system) will be implemented 3 days a week for 30 minutes in addition to the conventional rehabilitation program. Participants will receive a total of 4 weeks of treatment. Assessments will be made before initiating treatment, at the end of treatment, and 3 months after initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with unilateral or bilateral/triplegic spastic cerebral palsy
* Be between the ages of 5-15
* Levels I, II and III according to the Manual Ability Classification System (MACS)
* Have sufficient cognitive level, such as the ability to understand and follow simple instructions, and to perform desired tasks
* The upper extremity dimensions are suitable for the robot
* Parents and patients aged ≥ 9 years have agreed to participate in the study

Exclusion Criteria:

* Injection of antispasticity drugs (eg Botox) into upper extremity muscles and/or upper extremity orthopedic surgery in the last 6 months
* Having musculoskeletal disorders and peripheral nervous system disorders that impair the ability to use the upper extremity robotic system
* Having severe muscle spasticity and/or contracture
* Having uncontrolled seizures and/or presence of visually induced seizures
* Having severe learning difficulties, behavioral problems, skin lesions, visual and/or hearing difficulties that may affect function and participation

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-11-15 (Estimated)

PRIMARY OUTCOMES:
QUEST (Quality of Upper Extremity Skills Test) | Change from baseline Quality of upper extremity skills test at 4 weeks and 3 months
  It is a test developed to measure upper extremity functions. It consists of 7 sub-headings including dissociated movements, grasping, weight bearing, protective extension, hand function rating, spasticity rating and cooperativeness rating.

SECONDARY OUTCOMES:
ABILHAND-Kids | Change from baseline ABILHAND-Kids at 4 weeks and 3 months
  It is a functional scale developed to measure manual abilities. It measures the child's manual ability during daily activities and parents are asked to evaluate during these activities. The test consists of 21 questions and parents answer the questions in the test as impossible, difficult or easy. It is scored as impossible: 0, difficult: 1, easy: 2. The maximum score in the test is 42 and the minimum score is 0. Higher scores indicate better manual ability.
Box and Block Test | Change from baseline Box and Block Test at 4 weeks and 3 months
  It is a time-based test that evaluates rough manual dexterity. The participant is asked to throw the cubes on one side of a wooden box divided into two into the other compartment, and the result is obtained by counting how many cubes he has thrown in 60 seconds.
KINDL (Questionnaire to assess Health-Related Quality of Life in children and adolescents) | Change from baseline KINDL at 4 weeks and 3 months
  It is a questionnaire that measures the quality of life in children and adolescents, and there are child and family forms for different age groups. In this study, KINDL 3-6 age family form and 7-17 age family form will be used. KINDL 3-6 age family form is a questionnaire consisting of 52 questions in total about physical well-being, emotional well-being, self-esteem, family, social relations, kindergarten/nursery, other questions and illness. KINDL 7-17 age family form is a questionnaire consisting of 30 questions in total about physical well-being, emotional well-being, self-esteem, family, social relations, school, and illness. Parents answer questions as never, rarely, sometimes, often, or always. Questions are scored from 1 to 5. Negative questions are scored by reversing. Each section is scored between 0-100. A higher score indicates a higher quality of life.
Modified Ashworth Scala (MAS) | Change from baseline Modified Ashworth Scala at 4 weeks and 3 months
  It is used to evaluate the severity of spasticity. The joint is moved passively throughout the range of motion and the felt resistance is evaluated. In this study, shoulder adductors, elbow flexors, wrist flexors, and finger flexors will be evaluated with MAS. Spasticity severity is evaluated in 4 degrees. (0: no increase in muscle tone, 4: affected parts are rigid in flexion and extension). Higher scores indicate greater spasticity severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)

REFERENCES:
- [Background] Chen YP, Howard AM. Effects of robotic therapy on upper-extremity function in children with cerebral palsy: A systematic review. Dev Neurorehabil. 2016;19(1):64-71. doi: 10.3109/17518423.2014.899648. Epub 2014 Apr 11. PMID 24724587
- [Background] Fasoli SE, Ladenheim B, Mast J, Krebs HI. New horizons for robot-assisted therapy in pediatrics. Am J Phys Med Rehabil. 2012 Nov;91(11 Suppl 3):S280-9. doi: 10.1097/PHM.0b013e31826bcff4. PMID 23080043